CLINICAL TRIAL: NCT00406094
Title: The Evaluation of Singulair for the Treatment of Non-Allergic Rhinitis Eosinophil Syndrome (NARES)
Brief Title: Singulair Use in Non-Allergic Rhinitis Eosinophil Syndrome (NARES)
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bernstein, Jonathan A., M.D. (Individual)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Jonathan A. Bernstein, MD, Bernstein Clinical Research Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NARES
Record Dates: First submitted 2006-11-30; First posted 2006-12-04 (Estimated); Last update posted 2009-01-16 (Estimated); Status verified 2009-01

CONDITIONS: Rhinitis
Keywords: NARES; eosinophils; nasal symptoms
MeSH Terms: conditions — Rhinitis | interventions — montelukast

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor

ARMS (2):
- 1 (Experimental): montelukast
  Interventions: Drug: montelukast
- 2 (Placebo Comparator): placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: montelukast — 10mg
  Other Names: Singulair
  Arms: 1
Drug: placebo — placebo
  Arms: 2

SUMMARY:
The purpose of this trial is to determine if patients with NARES treated with montelukast (Singulair) will have improved nasal symptom scores and reduced nasal eosinophils.

DETAILED DESCRIPTION:
Patients will receive either montelukast or placebo in the treatment of NARES. 4 visits will be conducted over 12 weeks. A history and physical will be performed at the beginning of the trial and at the end. Skin testing will be done at Visit 1. Nasal smears and lavages will be performed at every visit. Patients will be compensated for time and travel.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 - 65 years
* Diagnosed with NARES

Exclusion Criteria:

* Smokers, exposed to passive smoke
* Diagnosis of seasonal allergic rhinitis (SAR), perennial allergic rhinitis (PAR), or vasomotor rhinitis (VMR)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2006-11; Primary Completion 2009-12 (Estimated); Study Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
Determine whether montelukast is more effective than placebo at reducing the number of nasal eosinophils associated with NARES | December 2008
Determine whether montelukast is more effective than placebo at reducing nasal symptom scores | December 2008

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan A Bernstein, MD, Principal Investigator — Bernstein Allergy Group
Locations (1):
- Bernstein Allergy Group, Cincinnati, Ohio, United States